CLINICAL TRIAL: NCT00940433
Title: Four Arm Randomised Trial Comparing Laparoscopic And Open Hernia Repairs
Brief Title: Hernia Repair Four Arm Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Yasser Hamza, Faculty of Medicine, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: # 90713
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Inguinal Hernia
Keywords: Minimally invasive; Inguinal hernia; Pro-peritoneal repair
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetra-4-amidinophenoxypropane; tetraethylpyrazine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- open properitoneal (Active Comparator): patients undergoing open properitoneal hernia repair
  Interventions: Procedure: open properitoneal hernia repair
- Lechtenstien repair (Active Comparator): Patients undergoing Lechtestien hernia repair
  Interventions: Procedure: Lechtestien hernia repair
- Laparoscopic transperitoneal repair (Active Comparator): Patients undergoing TAPP repair
  Interventions: Procedure: Laparoscopic transperitoneal approach
- Lap totally extraperitoneal approach (Active Comparator): Patients undergoing TEP approach
  Interventions: Procedure: Laparoscopic totally extraperitoneal approach

INTERVENTIONS:
Procedure: open properitoneal hernia repair — suprapubic retro-inguinal approach
  Other Names: extraperitoneal repair
  Arms: open properitoneal
Procedure: Lechtestien hernia repair — onlay mesh repair
  Other Names: tension free repair
  Arms: Lechtenstien repair
Procedure: Laparoscopic transperitoneal approach — intraperitoneal insufflation followed by re-exiting to the hernia site
  Other Names: TAPP
  Arms: Laparoscopic transperitoneal repair
Procedure: Laparoscopic totally extraperitoneal approach — avoiding the peritoneum altogether
  Other Names: TEP
  Arms: Lap totally extraperitoneal approach

SUMMARY:
This study compares the outcome of the four most commonly used operations for the repair of primary groin hernia including the new key hole surgical techniques. It aims at answering the question of whether the new technology really improve the outcome, saves time and reduce patient suffering.

DETAILED DESCRIPTION:
The study compares two traditional techniques of inguinal hernia repair; namely Lechtenstien repair and properitoneal repair versus two techniques of laparoscopic hernia repair, namely extraperitoneal and transperitoneal repair. It compares the operative time, complications, postoperative pain and the speed of patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* adult male primary inguinal hernia

Exclusion Criteria:

* recurrent hernia previous lower abdominal surgery [excluding appendectomy]

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
patient ability to resume domestic activity independently | daily reporting by the patient

SECONDARY OUTCOMES:
time of the patient to return to work | reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Hamza, A professor, Principal Investigator — University of Alexandria
Locations (1):
- Main University hospital, Alexandria, Alexandria Governorate, Egypt